CLINICAL TRIAL: NCT06785272
Title: Magnesium Trial in Acute Asthma in Emergency Department
Acronym: MAGICIAN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzanne Schuh (Other)
Collaborators: Alberta Children's Hospital (Other); McMaster Children's Hospital (Other); Stollery Children's Hospital (Other); Children's Hospital of Eastern Ontario (Other); St. Justine's Hospital (Other); The Hospital for Sick Children (Other)
Responsible Party: Sponsor-Investigator, Suzanne Schuh, Staff Physician, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5274
Record Dates: First submitted 2025-01-09; First posted 2025-01-21 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Asthma
Keywords: asthma, magnesium sulfate; pediatric, acute asthma
MeSH Terms: conditions — Asthma | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): This group will receive a single dose of intravenous magnesium sulfate over 30 minutes. After this treatment has been completed, they may also get further Ventolin inhalations or other asthma medicines which are not part of the study, as recommended by the emergency physician. The participant will be monitored closely by the study nurse who will measure their breathing, heart rate, blood pressure and oxygen for 3 hours after the study treatment. The study nurse will also notify the emergency physician of any major changes.
  Interventions: Drug: magnesium sulfate
- Placebo Group (Placebo Comparator): This group, will receive a single dose of intravenous placebo (normal saline, i.e. salt water) over 30 minutes. After this treatment has been completed, they may also get further Ventolin inhalations or other asthma medicines which are not part of the study, as recommended by the emergency physician who is taking care of the participant. They will be monitored closely by the study nurse who will measure the participant's breathing, heart rate, blood pressure and oxygen for 3 hours after the study treatment. The study nurse will also notify the emergency physician of any major changes in their health.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: magnesium sulfate — After initial therapy with the systemic CSs routinely used for acute asthma management at a given site, 3 treatments with inhaled salbutamol and ipratropium, eligible patients with PRAM ≥5 will, under the care of the research nurse, receive a 30-minute IV infusion of 75 mg/kg of Mg sulfate(maximum 2.0 g) [experimental group]
  Arms: Experimental Group
Drug: Normal Saline — After initial therapy with the systemic CSs routinely used for acute asthma management at a given site, 3 treatments with inhaled salbutamol and ipratropium, eligible patients with PRAM ≥5 will, under the care of the research nurse, receive a 30-minute IV infusion of 0.9% saline [control group].
  Arms: Placebo Group

SUMMARY:
Despite optimal initial emergency department (ED) therapy, 50% of children with severe acute asthma have ongoing moderate-severe respiratory distress. Guidelines recommend intravenous magnesium (IVMg) for them, yet evidence for IVMg efficacy is scant and disparate. While early small Randomized Controlled Trials (RCTs) suggested hospitalization benefit, recent large observational studies found no association between IVMg and improved outcomes. IVMg therapy is resource-intensive, can cause hypotension and demands close monitoring. Previous RCTs only assessed early Mg effect at 1-2 hours, overlooked the peak effect of key co-interventions such as corticosteroids and did not use validated scores. IVMg use is variable and often delayed until ≥4 hours after ED therapy is started and after the hospitalization decision has been made. Thus, in observational studies children given IVMg are 6-10 times more likely to be hospitalized; these studies have major confounding and the true IVMg treatment effect is thus unknown. To conclusively determine if IVMg alters the exacerbation course, it must be given early, and the primary outcome measure should be the severity of respiratory distress measured at the peak effect of key co-interventions to focus on a clinically meaningful and objective effect. The Pediatric Respiratory Assessment Measure (PRAM)-a valid, discriminative, reproducible and responsive-to-change instrument-is thus the ideal primary outcome measure. Hospitalization outcome has major confounding by indication and MD perceptions.

Primary Aim: In children with acute asthma remaining in moderate-severe distress after 1 hour of initial ED therapy, is early IVMg therapy associated with a significantly greater improvement in respiratory distress, measured by PRAM, at 2 hours after starting the intervention, compared to placebo? Hypothesis: IVMg will yield significantly greater PRAM improvement of ≥1.0 point than placebo.

Expected Outcomes: This trial will clarify if there is an incremental benefit of IVMg in decreasing respiratory distress in pediatric refractory acute asthma. A positive result will establish a proven standard of care for this indication, with a need for Knowledge Translation (KT) to implement routine early IVMg therapy. A negative result will lead to de-implementation of IVMg which may also lead to cost savings.

DETAILED DESCRIPTION:
The investigators propose a 6-centre randomized, double-blind, placebo-controlled trial. Two groups will be compared: IV Mg sulfate and IV (intravenous) 0.9% saline placebo. After initial therapy with the systemic Corticosteroids (CSs) routinely used for acute asthma management at a given site, 3 treatments with inhaled salbutamol and ipratropium (ipratropium use as per local practice), eligible patients with PRAM ≥5 will, under the care of the research nurse, receive a 30-minute IV infusion of 75 mg/kg of Mg sulfate (maximum 2.0 g) [experimental group] or an identical volume of 0.9% saline [control group]. Outcomes will be measured during the 180-minute observational period in the ED and at 72 hours post ED discharge.

ELIGIBILITY:
Inclusion criteria:

1. Age 2.00-17.99 years (prior to 18th birthday),
2. Diagnosis of asthma, defined as an asthma or probable asthma diagnosis/asthma-like phenotype made by a physician (this includes ED physician) in a patient who in the opinion of the treating ED physician requires therapy for acute asthma in the ED (GINA asthma guidelines, 2024).
3. Moderate-severe asthma after initial therapy with 3 treatments of inhaled salbutamol and ipratropium, defined as an eligibility PRAM ≥5, indicating a strong association with hospitalization.

Exclusion criteria:

1. Receipt of IVMg within 24 hours prior to ED arrival.
2. Need for airway support on arrival. (Airway support on arrival meeting exclusion criteria will include immediate need for high flow nasal cannula therapy, non-invasive CPAP/bi-PAP ventilation or invasive ventilation with endotracheal intubation, as decided by the attending Emergency Department (ED) physician. Supplemental oxygen therapy will not represent an exclusion criterion.)
3. Known renal, chronic pulmonary, neurologic, cardiac or systemic disease: these may influence outcomes after Mg.
4. Known hypersensitivity to Mg sulfate.
5. Previous enrollment.
6. Poor mastery of English and/or French language precluding informed consent understanding.
7. No phone/email; unavailable for follow-up

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Pediatric Respiratory Assessment Measure (PRAM) score: This score ranges from 0-12. A score from 0-3 is mild, 4-7 moderate and 8-12 severe. A low score is a better outcome and a high score is a worse outcome. | The primary outcome measure will be the PRAM score at 120 minutes post start of experimental therapy.
  PRAM is a validated 12-point asthma severity score which exhibits the most comprehensive measurement properties of all asthma scores and has been successfully used as an outcome in major trials. It is the only score with demonstrated criterion validity, using respiratory resistance as the gold standard. PRAM has been validated in both preschool and school-aged children in the ED with asthma and has strong association with admission. PRAM has inter-rater reliability above 70% and is adopted in all pediatric EDs in Canada. Most children treated for acute asthma are preschoolers who lack coordination to perform pulmonary function tests reliably. To maximize the accuracy of the PRAM measurement, all study nurses will complete an online PRAM training module. We will use an eligibility cut-off of PRAM ≥ 5 post initial therapy as this is associated with clinically concerning respiratory distress requiring further intervention. A PRAM score from 0-3 is mild, 4-7 moderate and 8-12 severe.

SECONDARY OUTCOMES:
Changes in PRAM score | Changes in PRAM score from baseline (pre intervention) to 30, 60, 120, 180 minutes after start of experimental therapy
  Changes in vital signs
Hospitalization for asthma at the index ED visit | Up to 24 hours after starting experimental therapy
  Defined as admission to an inpatient unit due to continued/worsening distress
Changes in respiratory rate | From baseline (pre-intervention) to 30,60,120 and 180 minutes post intervention (respiratory rate )
  Changes in vital signs
Changes in oxygen saturation | From baseline (pre-intervention) to 30,60,120 and 180 minutes post intervention ( oxygen saturation)
  Changes in vital signs
Changes in blood pressure | From baseline (pre-intervention) to 10,20,30,60,120, and 180 minutes post intervention (blood pressure).
  Changes in vital signs
PRAM denoting mild asthma (≤ 3 points is a widely accepted discharge criterion). | at 120 minutes post intervention
  Pediatric Respiratory Assessment Measure (PRAM) is a valid clinical score assessing acute asthma severity in toddlers and teenages. Score ranges from 0 to 12 (mild to severe). A higher score is a more severe asthma measurement. A low score is a better outcome than a high score.
Hospitalization for asthma at any medical facility | within 72 hours post- ED discharge
  Defined as admission to an inpatient unit due to continued/worsening distress
Unscheduled asthma-related visits to any health care provider | within 72 hours post- ED discharge
  Family-initiated asthma-related medical visit
Hospital length of stay. | From presentation at the Emergency Department triage to the time of hospital discharge, up to 4 weeks.
  Length of stay is the duration of a hospital stay in hours

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Schuh, MD, Principal Investigator — The Hospital for Sick Children
Locations (6):
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Ontario
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU-Sainte Justine Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No